CLINICAL TRIAL: NCT06864429
Title: Efficacy of Catheter Ablation of Frequent Asymptomatic Idiopathic Premature Ventricular Complexes in Treating Latent Left Ventricular Systolic Dysfunction As Being Assessed by Speckle Tracking of LV Global Longitudinal Strain
Brief Title: Impact of Catheter Ablation of Frequent Premature Ventricular Complexes in Treating Subtle Left Cardiomyopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD102/2023
Record Dates: First submitted 2025-02-14; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-01

CONDITIONS: Premature Ventricular Complexes; Ventricular Arrhythmias
Keywords: catheter ablation; radiofrequency ablation; Premature ventricular complexes; global longitudinal strain; PVCs induced cardiomyopathy; Idiopathic PVCs; Speckle tracking
MeSH Terms: conditions — Ventricular Premature Complexes | interventions — Catheter Ablation

STUDY DESIGN:
Intervention Model Description: group B ( ablation arm), will be applied for radiofrequency catheter ablation of PVCs as a treatment strategy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (control arm) (No Intervention): Group A is the control arm that will be applied to the standard of care treatment which is follow-up of symptoms status and left ventricular ejection fraction as per the recommendation of ESC guidelines of management of ventricular arrhythmias and sudden cardiac death published in 2022.
- Group B (ablation arm) (Active Comparator): Group B is the ablation arm that will be scheduled for radiofrequency catheter ablation of PVCs.
  Interventions: Procedure: Radiofrequency catheter ablation

INTERVENTIONS:
Procedure: Radiofrequency catheter ablation — Radiofrequency (RF) catheter ablation is a minimally invasive procedure that targets and eliminates certain types of cardiac arrhythmias. RF became effective as the first-line treatment for ventricular arrhythmias in some circumstances.
  Arms: Group B (ablation arm)

SUMMARY:
Throughout the past decade, there were no straightforward recommendations regarding the management of asymptomatic high-burden Premature ventricular complexes (PVCs) in structurally normal heart extending from the European Society of Cardiology (ESC) guidelines of management of ventricular arrhythmias in 2014, passing by the American Heart Association (AHA), American College of Cardiology (ACC), and Heart Rhythm Association (HRA) guidelines 2017, and reaching to the recent ESC guidelines in 2022 that declared overtly that there is a gap of evidence regarding management of asymptomatic high burden PVCs in structurally normal heart.

The goal of this clinical trial is to know if other imaging modalities rather than the conventional Two-dimension (2D) echocardiography can guide the treatment strategy of high-burden idiopathic premature ventricular complexes (PVCs). In our clinical trial, we used 2D speckle tracking of left ventricular (LV) global longitudinal strain (GLS) as an indicator for subtle LV systolic dysfunction in patients with structurally normal heart by conventional echocardiography.

The main questions the trial aims to answer are:

* Is radiofrequency catheter ablation an effective method in the treatment of early subtle myocardial dysfunction in patients with normal left ventricle ejection fraction (LVEF) and internal dimensions guided by 2D STE of GLS before progression into overt LV systolic dysfunction?
* Is there a correlation between radiofrequency catheter ablation of asymptomatic frequent idiopathic PVCs and improvement of patient functional capacity as an indicator for subconscious adaptation?
* Is there a correlation between PVC burden and the degree of impairment of GLS?

Researchers will compare group A (control group) and group B (ablation group) to see if there is a significant difference between them regarding global longitudinal strain.

Participants will be randomized into two groups each containing 20 patients. Group A (Control group): will be subjected to the standard of care being regular follow-up of symptom status and left ventricular ejection fraction (LVEF) Group B (ablation group): will be scheduled for PVC ablation.

DETAILED DESCRIPTION:
The clinical trial was conducted from June 2023 to August 2024. A total of 218 patients entered the screening phase. Of that participant pool, 116 patients did not fulfill the eligibility criteria since 90 patients were symptomatic, 33 patients had more than one PVC morphology in Holter ECG monitoring, 10 patients had episodes of atrial fibrillation (AF) in Holter ECG monitoring, 2 patients were diagnosed with chronic obstructive pulmonary disease (COPD), 1 patient had chronic kidney disease (CKD).

The other 100 patients continued with the subsequent stage of assessment of LV GLS, as mentioned in the outlined methodology. Of this cohort, 60 patients were excluded from the study because they did not meet the criteria for randomization, as they showed normal LV GLS ≥ -16%.

Accordingly, our study was conducted on 40 patients meeting the inclusion criteria mentioned. Those patients were further randomized into two groups each containing 20 patients.

Group A (Control group): subjected to the standard of care being regular follow-up of symptom status and left ventricular ejection fraction (LVEF) Group B (ablation group): scheduled for PVC ablation.

After a minimum duration of 3 months all participants were applied to follow-up assessment of symptoms status, 6-minute walk test (6MWT), PVC burden by Holter ECG monitoring, LV GLS by speckle tracking Echocardiography (STE).

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic patients with frequent idiopathic PVCs, defined as PVCs burden of ≥ 20% of total beats in Holter ECG monitoring in the structurally normal heart as being assessed by conventional 2D echocardiography and normal 12 lead surface ECG.
* Impaired LV GLS by 2D speckle tracking (GLS > -16 %).
* Patients willing and capable of providing informed consent

Exclusion Criteria:

* Multiple co-morbidities that may be potential factors affecting functional capacity including anemia, Chronic obstructive pulmonary disease (COPD), interstitial pulmonary fibrosis, bronchial asthma, Cerebrovascular stroke (CVS), skeletomuscular abnormalities or chronic kidney disease (CKD).
* Symptoms including but not limited to fatigue, palpitations, dyspnea, chest pain, dizziness, syncope, presyncope, or functional limitation that was defined as less than the lower limit of predicted 6-minute walk distance (6 MWD).
* Any electrolyte abnormalities, abnormal arterial blood gases, and/or abnormal thyroid profile.
* Ischemic heart disease (ISHD), in our study ISHD was defined as patients with a previous history of Myocardial infarction, acute coronary syndrome, previous revascularization with percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG), or objective evidence of myocardial ischemia including noninvasive functional assessment or coronary angiography showing significant stenosis > 50%.
* Symptomatic or asymptomatic structural heart disease including any congenital heart diseases, significant valvular lesion defined as primary or secondary valvular lesion causing abnormal loading condition, or more than grade I diastolic dysfunction.
* Any symptomatic or asymptomatic phenotype of cardiomyopathies.
* Polymorphic PVCs.
* Atrial fibrillation.
* Positive family history of sudden cardiac death.
* Heart failure including heart failure with preserved ejection fraction (HFpEF), heart failure with mildly reduced ejection fraction (HFmrEF), and heart failure with reduced ejection fraction (HFrEF).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — male and female
Enrollment: 40 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
global longitudinal strain | minimum of 3 months after (intervention) radio frequency ablation
  change of left ventricular global longitudinal strain was an indicator of the effectiveness of radiofrequency ablation in the treatment of subtle LV systolic dysfunction and prevention of further progression into overt cardiomyopathy.

SECONDARY OUTCOMES:
functional capacity | minimum of 3 months after (intervention) radio frequency ablation
  The trial aims to assess the correlation between radiofrequency catheter ablation of asymptomatic frequent idiopathic PVCs and change of patient functional capacity that is evaluated by a 6-minute walk test as an indicator for subconscious adaptation
PVC burden | minimum of 3 months after (intervention) radio frequency ablation
  The trial aims to assess the correlation between PVC burden and the degree of impairment of GLS

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university hospital, Cairo, Abbasya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided